CLINICAL TRIAL: NCT00991003
Title: A New Method for Colorectal Cancer Screening: Colon Capsule Endoscopy Compared to Conventional Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Julia Pilz, Resident, University Hospital Basel, Gastroenterology, University Hospital Basel
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: EKBB25407
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2009-10-07 (Estimated); Status verified 2009-10

CONDITIONS: Colorectal Cancer
Keywords: Colon Capsule Endoscopy; Colorectal Cancer; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Colon capsule endoscopy and colonoscopy (Experimental): Patients underwent CCE on day 1 and conventional colonoscopy on day 2
  Interventions: Procedure: Colon capsule endoscopy; Procedure: Conventional Colonoscopy

INTERVENTIONS:
Procedure: Colon capsule endoscopy — The PillCam® Colon Capsule is 11mm x 31mm in size (Figure 1), is equipped with two cameras acquiring pictures from both ends of the capsule at a rate of 4 frames per second (2 pictures per second and camera). The PillCam® Colon Capsule is automatically activated when it is removed from the package. It enters sleeping mode after approximately 10 minutes and starts transmitting again 1 h 45 min later. It has a total operating time of 8 - 10 hours. During the examination the patient wears a sensor array which is attached to the abdominal skin and a data recorder for storage of the information generated by the ingested capsule. After the examination the data are downloaded into the Given Imaging workstation and a video is generated.
  Other Names: Pillcam Colon Capsule
Procedure: Conventional Colonoscopy

SUMMARY:
Introduction:

Prevention of colorectal cancer (CRC) is feasible through polypectomy on screening colonoscopy. Patient acceptance remains the main limiting factor for execution. Colon capsule endoscopy (CCE) might be a novel method for large populations.

Aims and methods:

Patients referred for screening means or lower gastrointestinal complaints were included in this single center pilot study. They underwent preparation and then ingested the capsule (PillCam Colon). Standard colonoscopy was performed the next morning. Significance was defined as polyps >5mm in size. Performance of exams was by independent physician with blinding of results.

DETAILED DESCRIPTION:
Study design This was a prospective, single center pilot analysis under screening conditions. Patient enrollment was from November 5, 2007, to May 7, 2008. All patients provided written informed consent. Patients underwent CCE on day 1 and conventional colonoscopy on day 2, the examinations were done by different physicians. Results were blinded until both examinations had been completed and until interobserver evaluation was finished. Patient acceptance was assessed with a questionnaire after completion of both examinations.

This study was approved by the ethics committee. The study was partly funded by the Nycomed Fund of the University Hospital Basel, Switzerland and by Given Imaging Ltd., Yoqneam, Israel).

The authors designed the study, gathered and analyzed the data; the sponsors had no role in design or conduct of the study nor did they review or approve the data.

Patients Men and women above the age of 50 years without symptoms (Indication for screening) or with lower gastrointestinal signs and symptoms and individuals younger than 50 years, minimum 18 years, without symptoms but with a positive family history for colorectal cancer (CRC) (Indication for screening) were considered for this study. Exclusion criteria were CRC in the patient's history, cardiac pacemaker, contraindications for sodium phosphate solution (Colophos®) and risk factors for capsule retention including surgical intestinal anastomosis, Crohn's disease, diverticulitis and radiologically suspected bowel obstruction.

Data collection General characteristic of the patients were assembled, including demographics, family history and recent surgery, as well as bowel habits.

Hypothesis, Aim and End Points Significance was defined as polyps >5mm in size, with the hypothesis that detection rate on CCE corresponds with colonoscopy. The aim was to evaluate a novel method (colon capsule endoscopy) for performance as a screening tool compared to conventional colonoscopy in asymptomatic patients. The proclaimed benefit would be an increase in acceptance of screening for colorectal cancer and a probable better detection rate of adenoma resp. carcinoma.

The primary endpoint was the number of cancerous lesions and polyps detected on CCE compared to conventional colonoscopy. Secondary endpoints were completeness of the exam completeness, patient acceptance and adherence to preparation regimen.

Colon preparation and Propulsion of the Capsule For colon cleansing we applied our department's standard preparation procedure for conventional colonoscopy including diet and Macrogolum (PEG, Cololyt®; Spirig Pharma, Egerkingen, Switzerland) and added an oral motility agent, Phospho Soda (Colophos®; Spirig Pharma, Egerkingen, Switzerland)-boosters and a rectal suppository that promotes defecation, Table 1. Patients started with a low residual diet three days prior to the PillCam® Colon examination. The following day they were required to adhere to a liquid diet and one day before the examination to a clear liquid diet. The evening before the examination they ingested 2 litres of Cololyt® between 18:00 and 19:30 and continued with another 2 litres the next morning between 7:00 and 8:30. At 11:00 they were given 2 tablets of Domperidon (Motilium®; Janssen-Cilag AG, Baar, Switzerland) 10mg a couple of minutes prior to the PillCam® Colon capsule. Propulsion from stomach to small bowel was verified using real time viewing before giving the first Colophos® booster (45 ml). That we later abandoned (for the remaining 49 patients) due to satisfactory propulsion. If the capsule had not been excreted by 17:00 (3 hours after the first dose) a second dose of 30 ml Colophos® was added. If it still had not been excreted by 19:30, a suppository of Bisacodylum 10 mg (Prontolax®; Streuli Pharma, Uznach, Switzerland) was administered. The patient removed electrodes and recorder-belt at the excretion of the capsule or at 22:00, which ever came first, and continued clear liquid diet until the conventional colonoscopy was performed the following day.

Pillcam Colon Capsule The PillCam® Colon Capsule is 11mm x 31mm in size (Figure 1). It is equipped with two cameras acquiring pictures from both ends of the capsule at a rate of 4 frames per second (2 pictures per second and camera). Compared to the PillCam® Small Bowel capsule the optic is optimized and more than double of the area coverage and depth view are provided. The PillCam® Colon Capsule is automatically activated when it is removed from the package. It enters sleeping mode in order to save energy after approximately 10 minutes and starts transmitting again 1 h 45 min later. It has a total operating time of 8 - 10 hours. During the examination the patient wears a sensor array which is attached to the abdominal skin and a data recorder for storage of the information generated by the ingested capsule. After the examination the data are downloaded into the Given Imaging workstation and a video is generated.

ELIGIBILITY:
Inclusion Criteria:

* male/female above the age of 50 years with symptoms (Indication for screening)
* male/female above the age of 50 years without symptoms
* male/female younger than 50 years without symptoms but with a positive family history for colorectal cancer (CRC) (Indication for screening)

Exclusion Criteria:

* CRC in the patient's history
* cardiac pacemaker
* contraindications for sodium phosphate solution (Colophos®)
* risk factors for capsule retention including surgical intestinal anastomosis, Crohn's disease, diverticulitis and radiologically suspected bowel obstruction

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was the number of cancerous lesions and polyps detected on CCE compared to conventional colonoscopy | 7 Months

SECONDARY OUTCOMES:
Secondary endpoints were completeness of the exam completeness, patient acceptance and adherence to preparation regimen | 7 Months

CONTACTS AND LOCATIONS:
Overall Officials: Julia B Pilz, MD, Principal Investigator — University Hospital, Basel, Switzerland; Christoph Beglinger, MD, Study Director — University Hospital, Basel, Switzerland; Lukas Degen, MD, Study Chair — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Pilz JB, Portmann S, Peter S, Beglinger C, Degen L. Colon Capsule Endoscopy compared to Conventional Colonoscopy under routine screening conditions. BMC Gastroenterol. 2010 Jun 18;10:66. doi: 10.1186/1471-230X-10-66. PMID 20565828